CLINICAL TRIAL: NCT02855398
Title: Understanding Decision-Making and the Relationship to Food Intake in Children 7 to 11 Years Old
Brief Title: Decision-Making and the Relationship to Food Intake in Kids
Acronym: DMK
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Assistant Professor, Department of Nutritional Sciences and Food Science, Penn State University
Other Study IDs: DecisionMakingEatingKids01
Record Dates: First submitted 2016-06-29; First posted 2016-08-04 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this 18-month project is to investigate how decision-making influences food choice and consumption in children ages 7 to 11 years old. Although several studies suggest that the ability to make good decisions relates to eating behaviors, no studies have looked at how food reward influences the decision-making process to impact actual food intake. This proposal will answer these questions and bridge this gap in knowledge, which could lead to the development of more effective interventions for childhood obesity. To accomplish this, the investigators have assembled a diverse team with expertise in food intake, nutrition, and decision sciences. First, the investigators will establish if there are differences in decision-making between children varying in weight status. Second, the investigators will determine if performance on behavioral decision-making tasks relates to food consumption in the laboratory. Third, the investigators will examine response functional magnetic resonance imaging (fMRI) blood-oxygen-level-dependent (BOLD) response to various rewards (i.e. food and money) and determine if this is influenced by child weight status. Fourth, the investigators will examine differences in fMRI BOLD at rest in decision-making regions are correlated with food intake and weight status. Eighty-two children will participate in our study. The long-term goal of this project is to investigate if there are differences in brain regions corresponding to these behaviors in overweight children and if these differences relate to eating behaviors in this population. Children will undergo fMRI while playing a reward task as well as consume meals in our laboratory. Decision-making will also be assessed by having children complete various behavioral measurements of reward and inhibitory control.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* English as native language
* Reading at/above grade level
* Not Claustrophobic
* Generally Healthy

Exclusion Criteria:

* Left-handedness
* Metal in or on body that cannot be removed
* Claustrophobia
* Medication usage that may alter brain activity or blood flow
* Medical disorder that may impact comfort of safety in MRI scanner
* Food Allergies
* Dietary Restrictions
* Learning Disabilities
* Psychiatric Disorders

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 7-11 years old.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI), blood-oxygen-level-dependent (BOLD) response to various reward types (food, money, no reward). | Collected at fMRI scan at week 4
  Regions of interest BOLD analysis of an fMRI card-guessing task for various reward types
Functional magnetic resonance imaging (fMRI), blood-oxygen-level-dependent (BOLD) response at rest (resting-state fMRI) | Collected at fMRI scan at week 4
  Regions of interest BOLD analysis of resting-state fMRI to examine differences in brain regions of interest at rest
Behavioral inhibitory control task | Collected at either week 1-3 (randomized)
  Measured by performance on a go/nogo task
Behavioral reward inhibitory control task | Collected after the behavioral inhibitory control task (same visit), which is either week 1-3 (randomized)
  Measured by performance on a go/nogo task with a reward incentive
Behavioral risk-taking and reward task | Collected at either week 1-3 (randomized)
  Measured by performance on the hungry donkey task
Behavioral dietary self-control assessment | Collected at either week 1-3 (randomized)
  Measured by performance on a dietary self-control task

SECONDARY OUTCOMES:
Energy intake at baseline | Collected at either week 1-3 (randomized)
  Measured at an objective laboratory test-meal (kcal and grams)
Energy intake at a buffet meal | Collected at either week 1-3 (randomized)
  Measured at an objective laboratory test-meal (kcal and grams)
Energy intake after a meal preload | Collected at either week 1-3 (randomized) following the baseline meal
  Measured at an objective laboratory test-meal (kcal and grams)
Functional magnetic resonance imaging (fMRI), blood-oxygen-level-dependent (BOLD) response to various reward types (food, money, no reward). | Collected at week 4
  Whole brain BOLD analysis of an fMRI card-guessing task for various reward types
Functional magnetic resonance imaging (fMRI), blood-oxygen-level-dependent (BOLD) response at baseline | Collected at week 4
  Whole brain BOLD analysis of an fMRI card-guessing task for various reward types

OTHER OUTCOMES:
Liking of foods | Collected after each meal at multiple time points during weeks 1-4
  Ratings of how much the child likes each food in the meal on a visual analog scale
Fullness feelings | Collected at multiple time points during weeks 1-4
  Ratings of how full the child feels measured on a child-friendly visual analog scale
Pubertal Development | Collected at week 1
  Child report of pubertal status questionnaire
Height | Collected at week 1
  Height in cm measured by stadiometer
Weight | Collected at week 1
  Weight in kg measured by a standard digital scale
Body fat percentage | Collected at week 1
  Assessed by bioelectrical impedance analysis scale
Body mass index | Collected at week 1
  Calculated from height, age, sex
BMI percentile | Collected at week 1
  Calculated from height, weight, age and sex - according to the Center for Disease Control (CDC) standards
BMI z-score | Collected at week 1
  Calculated from height, weight, age and sex - according to CDC standards
Fat mass index | Collected at week 1
  Calculated from height, weight, age, sex
Fat-free mass index | Collected at week 1
  Calculated from height, weight, age, sex
Appetitive traits | Collected at week 1
  Parent-reported questionnaire of habitual eating styles in children
Parental feeding strategies | Collected at week 1
  Parent-reported questionnaire of feeding practices
Family demographics | Collected at week 1
  Parent-report questionnaire
Loss of control eating | Collected at week 4
  Loss of control when eating is frequently reported in middle childhood. Loss of control when eating was assessed via interview-style questionnaire to determine pre-clinical binge-like eating behaviors that may influence the primary outcome of energy intake at the 4 conditions of test-meals.
Inhibitory control and reward sensitivity questionnaires | Collected on either week 1-3 (randomized)
  Parent and child report of inhibitory control and reward sensitivity on a questionnaire
Age | Collected at the week 1
  Age of participant
Sex | collected at week 1
  sex of participant
Parent height | collected at week 1
  height in cm of parent measured by a stadiometer
Parent weight | collected at week 1
  weight in kg of parent measured by a standard digital scale
parent body fat | collected at week 1
  measured by bioelectrical impedance
Puberty Assessment Parental Report | Collected at week 1
  Parent report of pubertal status questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Shana Adise, B.S., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adise S, White CN, Roberts NJ, Geier CF, Keller KL. Children's inhibitory control abilities in the presence of rewards are related to weight status and eating in the absence of hunger. Appetite. 2021 Dec 1;167:105610. doi: 10.1016/j.appet.2021.105610. Epub 2021 Jul 26. PMID 34324909
- [Derived] Adise S, Geier CF, Roberts NJ, White CN, Keller KL. Is brain response to food rewards related to overeating? A test of the reward surfeit model of overeating in children. Appetite. 2018 Sep 1;128:167-179. doi: 10.1016/j.appet.2018.06.014. Epub 2018 Jun 8. PMID 29890186